CLINICAL TRIAL: NCT06359015
Title: Use of Combination Metformin and Esomeprazole in Preterm Pre-eclampsia: a Randomized Controlled Trial
Brief Title: Metformin and Esomeprazole in Preterm Pre-eclampsia
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Lost funding
Sponsor: Christiana Care Health Services (Other)
Responsible Party: Principal Investigator, Kendall Bielak, MD, Resident Physician, Christiana Care Health Services
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 41138; 605095 (Other: DDD)
Record Dates: First submitted 2024-03-30; First posted 2024-04-11 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Preeclampsia Severe; Pre-Eclampsia; Preeclampsia; Preeclampsia Second Trimester; Preeclampsia Complicating Childbirth; Preeclampsia Puerperium; Preterm
Keywords: Metformin; Esomeprazole; Preterm Preeclampsia; Preeclampsia with Severe Features; Superimposed Preeclampsia with Severe Features
MeSH Terms: conditions — Pre-Eclampsia; Premature Birth | interventions — Metformin; Esomeprazole

STUDY DESIGN:
Intervention Model Description: There are two groups: experimental and control. The control group receives expectant management. The experimental group receives expectant management and medication treatment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Metformin and Esomeprazole (Experimental): Patients diagnosed with preterm preeclampsia receive expectant management with additional metformin/esomeprazole.
  Interventions: Drug: Metformin; Drug: Esomeprazole
- No Intervention (No Intervention): Patients diagnosed with preterm preeclampsia receive expectant management only.

INTERVENTIONS:
Drug: Metformin — Oral Metformin schedule:
  Day 1: 500 milligrams in morning Day 2: 500 milligrams two times a day Day 3: 1000 milligrams in morning, 500 milligrams in evening Day 4 onwards: 1000 milligrams two times a day based on individual tolerance
  Oral Esomeprazole schedule:
  40 milligrams Oral Esomeprazole daily until delivery which can be tapered down to 20 milligrams daily based on individual tolerance.
  Arms: Metformin and Esomeprazole
Drug: Esomeprazole — 40 milligrams Oral Esomeprazole daily until delivery which can be tapered down to 20 milligrams daily based on individual tolerance.
  Arms: Metformin and Esomeprazole

SUMMARY:
The purpose of this study is to better understand diagnosis and treatment of preterm preeclampsia. Currently, there are limited laboratory tests that can be used to diagnosis preeclampsia. Additionally, there are few treatments for this condition. This clinical trial will explore treatment options, Metformin and Esomeprazole, as well as serum markers that could improve the diagnosis and treatment of preterm preeclampsia.

DETAILED DESCRIPTION:
BACKGROUND:

The pathophysiology of preeclampsia

To achieve normal vascular function during pregnancy, the placental vascular endothelium secretes vasoactive substances and growth factors, most notably vascular endothelial growth factor (VEGF), sFlt-1, placental growth factor (PlGF) and soluble endoglin (sEng). These substrates interact with maternal natural killer cells to promote remodeling of the uterine spiral arteries in order to create a uteroplacental interface. Circulating vasoconstrictors, such as Thromboxane A2, and vasodilators play an important role in regulating the vascular endothelium in response to the developing uteroplacental interface.

In patients with preeclampsia, however, trophoblast cells demonstrate insufficient invasion of the spiral arteries, leading to poor remodeling, narrow vessel diameter and high vascular resistance. The endothelial dysfunction occurs in two phases. In the first phase, defective placental trophoblastic invasion of the uterine spiral arteries occurs at 14-18 weeks of gestation. This dysfunctional invasion leads to poor uteroplacental blood flow and the release of antiangiogenic factors and vasoconstrictive substances in the second phase.

In Defense of Metformin, Esomeprazole

Lower sFlt1 levels were detected in placental villous explants from patients diagnosed with preterm preeclampsia and treated with metformin. Metformin downgraded endothelial cell secretion by 53% and placental cell secretion by 63%. Similarly, in a meta-analysis of patients on metformin for gestational diabetes (GDM), Kalafat and Sukur concluded that the use of metformin was associated with a reduced risk of preeclampsia (relative risk (RR): 0.56; 95% confidence interval (CI): 0.37-0.85; n = 1260 women)

A recent randomized controlled trial by Cluver et al included 180 women with preterm pre-eclampsia between 26+0 to 31+6 weeks' gestation undergoing expectant management: 90 were randomized to extended release metformin and 90 to placebo. Investigators found that extended release metformin (3g daily) can prolong gestation in women with preterm pre-eclampsia

In vitro studies show proton pump inhibitors decrease soluble fems like tyrosine kinase -1 (sFlt-1) and soluble endoglin and improve markers of endothelial dysfunction. Esomeprazole reduces blood pressure in a preeclampsia transgenic mouse model that overexpresses sFlt-1.

Combination metformin and esomeprazole has shown promise in the treatment of preeclampsia as both agents reduce placental and endothelial secretion of sFlt-1 and soluble endoglin, and reduce endothelial dysfunction. Kaitu'u-Lino et al found that combining metformin and esomeprazole was additive at reducing sFlt-1 secretion and expression of sFlt-1 e15a mRNA isoform in primary cytotrophoblast, placental explants and endothelial cells.

Safety of Metformin, Esomeprazole

Metformin is a biguanide that inhibits hepatic gluconeogenesis and glucose absorption and stimulates glucose uptake in peripheral tissues.

In one large trial, 751 women with GDM were randomly assigned to receive insulin therapy or metformin. Both groups experienced similar rates of a composite outcome of perinatal morbidity, consisting of neonatal hypoglycemia, respiratory distress, need for phototherapy, birth trauma, prematurity, and low Apgar scores. Additionally, five randomized clinical trials showed the safety of metformin as well as its efficiency in dealing with GDM compared with insulin. A meta-analysis by Gui et al. demonstrated that metformin was superior to insulin in reducing the incidence of preeclampsia.

Proton pump inhibitors (PPI) such as esomeprazole have long-term safety data in the treatment of gastric reflux in pregnancy. The Motherisk Program conducted a meta-analysis on use of PPIs in 593 pregnancies and showed no increase in risk of malformations. Furthermore, in a large cohort study from the Swedish Medical Birth Registry on 955 infants whose mothers used PPIs during pregnancy showed no difference in birth weights, rates of congenital malformations, perinatal death, or low Apgar scores.

ELIGIBILITY:
Inclusion Criteria:

* Women 18 years or older
* Women diagnosed with preeclampsia or preeclampsia with severe features or superimposed preeclampsia with chronic hypertension
* Candidates for expectant management and had no clinical indication for immediate delivery

Exclusion Criteria:

* Delivery within 48hr is highly likely
* Maternal or fetal compromise that necessitated immediate delivery
* Diabetes or gestational diabetes currently on metformin therapy
* Reflux disease or other conditions currently on esomeprazole
* Contraindications to metformin, esomeprazole
* Baseline creatinine >124 μmol/L
* Hypersensitivity to metformin or esomeprazole
* Current use of metformin or esomeprazole
* Metabolic acidosis
* Use of drugs that might interact with metformin (glyburide, furosemide, or cationic drugs)
* Multiple gestations

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 4 (Actual)
Dates: Start 2021-02-11 (Actual); Primary Completion 2025-05-08 (Actual); Study Completion 2025-05-08 (Actual)

PRIMARY OUTCOMES:
Mean plasma difference in sFlt-1 | Over the first 14 days after randomization and during the remainder of pregnancy, an average of 3-4 months
  sFlt-1 from serum samples

SECONDARY OUTCOMES:
Mean plasma difference in vascular endothelial growth factor (VEGF) | Over the first 14 days after randomization and during the remainder of pregnancy, an average of 3-4 months
  VEGF from serum samples
Mean plasma difference in placental growth factor (PIGF) | Over the first 14 days after randomization and during the remainder of pregnancy, an average of 3-4 months
  PIGF from serum samples
Mean plasma difference in soluble endoglin (sEng) | Over the first 14 days after randomization and during the remainder of pregnancy, an average of 3-4 months
  sENG from serum samples
sFlt-1:PIGF ratio | Over the first 14 days after randomization and during the remainder of pregnancy, an average of 3-4 months
  sFLT-1:PIGF from serum samples
Prolongation of gestation | Over the first 14 days after randomization and during the remainder of pregnancy, an average of 3-4 months
  Difference in time of expectant management between experimental and control group.

CONTACTS AND LOCATIONS:
Overall Officials: Derek Bowden, MA,CIP,CHRC, Study Director — ChristianaCare Institutional Review Board
Locations (1):
- Christianacare Health System, Newark, Delaware, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cluver CA, Hiscock R, Decloedt EH, Hall DR, Schell S, Mol BW, Brownfoot F, Kaitu'u-Lino TJ, Walker SP, Tong S. Use of metformin to prolong gestation in preterm pre-eclampsia: randomised, double blind, placebo controlled trial. BMJ. 2021 Sep 22;374:n2103. doi: 10.1136/bmj.n2103. PMID 34551918
- [Background] Kaitu'u-Lino TJ, Brownfoot FC, Beard S, Cannon P, Hastie R, Nguyen TV, Binder NK, Tong S, Hannan NJ. Combining metformin and esomeprazole is additive in reducing sFlt-1 secretion and decreasing endothelial dysfunction - implications for treating preeclampsia. PLoS One. 2018 Feb 21;13(2):e0188845. doi: 10.1371/journal.pone.0188845. eCollection 2018. PMID 29466360
- [Background] Rowan JA, Hague WM, Gao W, Battin MR, Moore MP; MiG Trial Investigators. Metformin versus insulin for the treatment of gestational diabetes. N Engl J Med. 2008 May 8;358(19):2003-15. doi: 10.1056/NEJMoa0707193. PMID 18463376